CLINICAL TRIAL: NCT03922529
Title: Modified Application of Cardiac Rehabilitation for Older Adults
Acronym: MACRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Forman, MD (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Washington University School of Medicine (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Daniel Forman, MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY20080044; 1R01AG060499-01 (NIH)
Record Dates: First submitted 2019-04-15; First posted 2019-04-22 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Cardiac Rehabilitation; Transition of Care
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: There will be two intervention groups 1) MACRO-I in which the research team will work with the participant and providers to facilitate CR; 2) Usual care as determined by their clinical providers.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Key investigators and well as the outcomes assessor at each site will remain blinded to participant group placement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Care after an acute heart event will be at the discretion of the participants' clinical providers.
  Interventions: Other: Usual Care
- MACRO-I (Experimental): A coaching intervention that supplements usual care.
  Interventions: Behavioral: MACRO-I

INTERVENTIONS:
Behavioral: MACRO-I — MACRO-I coaches engage with patients regularly while they are still inpatients, and then by telephone once they are discharged. Coaching incorporates innovative techniques for holistic risk assessment (medical, functional, psychosocial), guidance to initiate CR in a format aligned with each patient's risks and preferences (i.e., CR as either site-based, home-based, or in a hybrid format [site transitioning to home]), behavioral prompts based on their personal goals of care, and de-prescribing of sedating medications.
  Arms: MACRO-I
Other: Usual Care — Participants will receive usual care that is recommended by their providers. MACRO study personnel will follow the participant for the course of the study to assess endpoints in comparison to the MACRO-I arm.
  Arms: Usual Care

SUMMARY:
Modified Application of Cardiac Rehabilitation for Older Adults (MACRO) responds to a critical underuse of cardiac rehabilitation in older adults with a coaching model that addresses issues related to aging as a means to better facilitate cardiac rehabilitation (CR). MACRO is a randomized controlled trial (RCT) in which older adults with a CVD event are randomized between a MACRO intervention (MACRO-I) versus usual care. The MACRO-I is designed to facilitate CR as a means to augment functional recovery.

DETAILED DESCRIPTION:
This is a pragmatic RCT of 350 older adults eligible for CR: hospitalized adults aged ≥70 years with a primary diagnosis of acute myocardial infarction/ acute coronary syndrome, stable ischemic heart disease, revascularization (coronary artery bypass graft surgery, percutaneous coronary intervention), valvular heart disease (surgical or transcatheter valve replacement or repair), heart failure (with reduced or preserved ejection fraction) or peripheral arterial disease. Participants who consent to participate will be randomly assigned to a MACRO-intervention (MACRO-I) versus usual care. In the MACRO-I arm, participants receive coaching that incorporates innovative features designed to address needs of older adults. These include holistic risk assessment (medical, functional, psychosocial), guidance to facilitate CR in a format that aligns with each patient's own risks as well as their preferences (i.e., CR formatted as either site-based, home-based, or in a hybrid format [site transitioning to home]), behavioral reinforcements to promote CR based on their goals of care, and deprescribing of sedating medications. While usual care may include CR, it provides no coaching, and none of the innovations associated with MACRO-I coaching. Endpoints focus particularly on functional capacity achieved by improved implementation of CR.

Aim 1: To establish efficacy, safety, and acceptability of the MACRO-I via a RCT.

We hypothesize that after 3 months, compared to usual care, participants randomized into MACRO-I will have:

H1.1: Greater improvements in function as measured by Activity Measure for Post-Acute Care Computer Adaptive Test (AM-PAC-CAT) Basic Mobility Domain (3 month changes; primary outcome).

H1.2: Greater improvements in function as measured by AM-PAC CAT daily activity domain; accelerometry; depression; frailty; self-efficacy; quality of life.

H1.3: Greater CR participation and adherence. H1.4: Greater impact on readmissions and hospitalization.

Aim 2: To examine the durability of benefit of MACRO-I compared to usual care.

We hypothesize that after 6 and 12 months (12 months will be captured as timing allows), compared to usual care, participants randomized into MACRO-I will have:

H2.1: Greater improvement in AM-PAC-CAT basic mobility and daily activity domains; accelerometry; depression; frailty; self-efficacy; quality of life.

H2.2: Greater impact in readmissions and hospitalization at 6 and 12 months (12 months will be captured as timing allows).

Aim 3: To explore characteristics of patients who benefit the most from the MACRO-I as compared to usual care.

H3.1: We anticipate functional capacity and other baseline characteristics will identify those who benefit from the MACRO-I (exploratory).

The MACRO study originally began recruitment with a target sample size of N=480 in November 2019. The primary outcome measure at this time was the Short Physical Performance Battery (SPPB), and a battery of secondary outcome measures included assessments of hand grip strength, accelerometry, cognition, depression, health literacy, frailty, physical activity, nutrition, readiness for change, self efficacy, and quality of life. However, the COVID-19 pandemic disrupted the original MACRO protocol. In March 2020 per Data Safety and Monitoring Board (DSMB) decision, all study participants who were enrolled at that time were withdrawn and the study was suspended to address safety concerns of face-to-face assessments during the height of the pandemic. It was necessary to modify the protocol so it could administered fully remotely, without changing the original aims and innovation of the intervention.

The SPPB was no longer feasible or safe as a primary outcome measure, so the study team selected the Activity Measure for Post-Acute Care with Computerized Adaptive Testing (AM-PAC CAT). The AM-PAC CAT is used to measure self-reported daily activity, can reliably be used to detect change over time, and can be administered over the phone. It was determined that with this new outcome measure, a target sample size of N=374 would be sufficient to retain the same statistical power for the new primary outcome as the original protocol, assuming 80% retention. The secondary outcome assessments were also revised, changing to measures that could be administered remotely when needed and leaving in-person assessments optional contingent on COVID risk.

Following all regulatory approvals of the revised protocol and outcome measures, the study restarted recruitment in September 2020. Enrollment concluded in August 2023 after 416 participants had been consented and 350 randomized. The retention rate was higher than anticipated at 87.7% completion of the primary outcome measure at 3 months, which allowed for the same amount of power with a smaller sample size.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 year
* Eligible cardiovascular disease (CVD) diagnosis (hospitalization for acute myocardial infarction/ acute coronary syndrome, stable ischemic heart disease, revascularization (coronary artery bypass graft surgery and percutaneous coronary intervention, valvular heart disease (surgical or transcatheter replacements or repair for mitral regurgitation or aortic stenosis),heart failure (exacerbation or new diagnosis)
* English speaking
* Able to provide written informed consent
* Able to be assessed and undergo study interventions

Exclusion Criteria:

* Unstable medical condition as indicated by history, physical exam, and/or laboratory findings
* Presence of non-CVD conditions likely to be fatal within 12 months (e.g., metastatic cancer)
* Severe cognitive impairment: Short Blessed screening with a score of 13 or greater cannot consent (as indicated by medical record)
* Long-term care resident at admission with no plans to return to independent living
* Unable to participate in follow-up assessments by telephone or in person

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 416 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Forman, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Washington University in St. Louis, St Louis, Missouri
  - VA Pittsburgh Healthcare system, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The original recruitment target was 480 beginning in November 2019. Due to the COVID-19 pandemic, the DSMB recommended suspension and withdrawal of all enrolled subjects in March 2020. The protocol was revised to be fully remote, and recruitment was reinitiated with a smaller target sample in September 2020. Enrollment ended in August 2023. 416 subjects consented to the study (total enrolled), and 350 completed the required baseline assessments to be randomized to an intervention group.
Pre-assignment Details: After informed consent, subjects completed a set of baseline questionnaires. Participants who did not meet the score requirements on the Short Blessed cognitive assessment at baseline were disqualified before randomization. Other reasons for withdrawal prior to randomization assignment included subject-initiated withdrawal, adverse event, death, or loss to follow-up after discharge from inpatient hospital admission. Participants must have completed baseline assessments in order to be randomized.
Period: Overall Study
Arm/Group | MACRO-I | Usual Care
Started | 176 | 174
Completed | 140 | 131
Not Completed | 36 | 43
Not completed — Withdrawal by Subject | 13 | 12
Not completed — Death | 7 | 12
Not completed — Lost to Follow-up | 12 | 19
Not completed — Adverse Event | 1 | 0
Not completed — Death after withdrawal | 1 | 0
Not completed — Participant was contacted for final visit and declined to complete | 1 | 0
Not completed — Moved to assisted living and was unreachable for follow-up assessments | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants who completed the required baseline measures to be randomized to an intervention group. Participants who consented but were withdrawn or disqualified prior to randomization are not included.
Groups:
- Total: Total of all reporting groups
Arm/Group | MACRO-I | Usual Care | Total
Number analyzed (Participants) | 176 | 174 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years was collected at baseline as part of a demographic questionnaire. The mean age per intervention group is reported.
  years | 75.9 (4.9) | 76.4 (5.7) | 76.1 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex was collected on the baseline demographics questionnaire. It is reported as the frequency count per group.
  Participants
    Female | 50 | 58 | 108
    Male | 126 | 116 | 242
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was collected on the baseline demographics questionnaire. It is reported as the frequency count of participants per group.
  Participants
    Hispanic or Latino | 1 | 0 | 1
    Not Hispanic or Latino | 173 | 171 | 344
    Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was collected on the baseline demographics questionnaire (select all that apply). It is reported as the frequency count per group.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 18 | 21 | 39
    White | 155 | 152 | 307
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 176 | 174 | 350
Marital Status [Count of Participants; unit: Participants] — Marital status was collected on the baseline demographics questionnaire. It is reported as the frequency count of participants per group.
  Participants
    Married or permanent partnership | 95 | 102 | 197
    Widowed | 42 | 37 | 79
    Divorced or separated | 26 | 23 | 49
    Never married | 10 | 10 | 20
    In a relationship | 2 | 1 | 3
    Other | 1 | 1 | 2
Social Support [Count of Participants; unit: Participants] — Participants were asked on the baseline demographics survey whether they lived alone or with others. The number of participants in each group who responded that they lived alone, and the number of participants in each group who responded that they lived with others is reported as the count of participants and the percentage of participants out of the total number in each group.
  Participants
    Lives alone | 69 | 50 | 119
    Lives with others | 107 | 124 | 231
AM-PAC CAT [Mean (Standard Deviation); unit: score on a scale] — The AM-PAC-CAT is a self-reported activity limitations measure that assesses perceived difficulty and level of assistance/limitations (Basic Mobility Domain).
  The Basic Mobility domain characterizes basic movement and physical functioning activities, such as bending, walking, carrying, and climbing stairs. Scaled scores range from 0-104.9 with higher scores indicating greater activity levels/fewer limitations.
  The Daily Activity domain characterizes difficulty of daily activities. Scaled scores range from 0-115.4 with higher scores indicating greater activity levels/fewer limitations.
  score on a scale
    Basic Mobility | 57.3 (6.5) | 56.3 (7.4) | 56.8 (7.0)
    Daily Activity | 54.6 (8.6) | 55.2 (9.1) | 54.9 (8.8)
Average total active time/24 hours (minutes) [Mean (Standard Deviation); unit: minutes/24 hours] — Change in lifestyle physical activity will be measured by wrist worn accelerometry to assess change in movement. An index of average total active minutes (≥18mg) per 24 hour period will be prioritized to quantify physical activity volume. It is assumed that higher total active time represents a better outcome.
  minutes/24 hours | 324.1 (127.4) | 347.8 (130.0) | 335.0 (128.8)
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: score on a scale] — The PHQ-9 is a standardized and validated 9 item depression scale. Scores range from 0-27 points on the scale, with the higher score showing a greater possibility of depression.
  score on a scale | 4.7 (3.1) | 4.9 (2.8) | 4.8 (3.0)
Morley Frail Scale [Mean (Standard Deviation); unit: score on a scale] — The Frail Scale is a 5-item assessment of fatigue, resistance, ambulation, illnesses, and loss of weight. Scores range from 0-5 with a higher number indicating greater frailty.
  score on a scale | 2.3 (1.4) | 2.2 (1.4) | 2.2 (1.4)
Sullivan Cardiac Self Efficacy [Mean (Standard Deviation); unit: score on a scale] — The Sullivan Cardiac Self-Efficacy scale evaluates an individuals confidence to take care of themselves in association to their cardiac disease. It is scored on scale of 0 to 52 points, with a higher score indicating higher confidence.
  score on a scale | 34.8 (7.6) | 35.0 (7.2) | 34.9 (7.4)
Veterans RAND-12 [Mean (Standard Deviation); unit: score on a scale] — The Veterans RAND-12 is a short standardized and validated questionnaire evaluating quality of life. The 12 items are summarized into two scores, a "Physical Health Summary Measure {PCS-physical component score}" and a "Mental Health Summary Measure {MCS-mental component score}". Both scores range from 0 to 100 with a population mean of 50. These provide an important contrast between physical and psychological health status. A higher score indicates better physical or mental health, respectively.
  score on a scale
    Physical Summary Score | 28.6 (10.1) | 28.5 (10.4) | 28.5 (10.3)
    Mental Summary Score | 50.0 (10.0) | 49.8 (8.9) | 49.9 (9.5)
Modified Rapid Eating Assessment for Participants-Shortened Version [Mean (Standard Deviation); unit: score on a scale] — The modified REAP-S is a self-reported 17-item questionnaire used to assess eating habits. The overall summary score ranges from 17 to 53 points, with a higher score representing healthier dietary patterns.
  A modified version of the questionnaire was used for this project after receiving approval by the developers of the instrument.
  score on a scale | 31.1 (3.9) | 31.4 (4.3) | 31.2 (4.1)
Duke Activity Status Index [Mean (Standard Deviation); unit: score on a scale] — The Duke Activity Status Index (DASI) is a self-reported 12-item scale that has been validated in cardiac patients against peak VO2 and has been demonstrated to be a reliable and responsive tool to quantify physical activity in daily living. Scaled scores range from 0 to 58.2 points, with a higher score corresponding to a higher estimated functional capacity.
  score on a scale | 25.3 (15.7) | 25.6 (16.5) | 25.4 (16.1)
Fall History [Count of Participants; unit: Participants] — The frequency count of participants who self-reported that they had experienced one or more falls in the past 3 months at the time of the baseline assessment.
  Participants | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: AM-PAC-CAT - Basic Mobility Domain
Description: AM-PAC-CAT is a self-reported activity limitations measure that assesses perceived difficulty and level of assistance/limitations (Basic Mobility Domain). The Basic Mobility domain characterizes basic movement and physical functioning activities, such as bending, walking, carrying, and climbing stairs. Scaled scores range from 0-104.9 with higher scores indicating greater activity levels/fewer limitations.
Time Frame: 3 months, i.e., Baseline to 3-month change
Population: All 350 randomized participants were analyzed with multiple imputation (Markov Chain Monte Carlo or MCMC method) for any missing or incomplete outcomes data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 5.1 (7.5) | 5.0 (5.4)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.5430, Mixed Models Analysis; Adjusted for baseline value of the outcome as a covariate using linear mixed models and multiple imputation for missing data; Mean Difference (Final Values) = 0.5, Standard Error of Mean 0.8 — The adjusted difference from a model may not necessarily match the raw difference between groups

2. Secondary Outcome: AM-PAC-CAT - Basic Mobility Domain
Description: as for outcome 1
Time Frame: Baseline to 6-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 4.9 (6.7) | 5.2 (5.9)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.7625, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.2, Standard Error of Mean 0.8 — The adjusted difference from a model may not necessarily match the raw difference between groups

3. Secondary Outcome: AM-PAC-CAT - Basic Mobility Domain
Description: as for outcome 1
Time Frame: Baseline to 12-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 4.9 (7.3) | 5.3 (6.5)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.8842, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.1, Standard Error of Mean 0.7 — The adjusted difference from a model may not necessarily match the raw difference between groups

4. Secondary Outcome: AM-PAC-CAT - Daily Activity Domain
Description: AM-PAC-CAT is a self-reported activity limitations measure that assesses perceived difficulty and level of assistance/limitations (Basic Mobility Domain). The Daily Activity domain characterizes difficulty of daily activities. Scaled scores range from 0-115.4 with higher scores indicating greater activity levels/fewer limitations.
Time Frame: Baseline to 3-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 5.8 (8.8) | 4.5 (11.1)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.4086, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.0, Standard Error of Mean 1.2 — The adjusted difference from a model may not necessarily match the raw difference between groups

5. Secondary Outcome: AM-PAC-CAT - Daily Activity Domain
Description: as for outcome 4
Time Frame: Baseline to 6-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 6.3 (10.0) | 5.2 (10.6)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.3841, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.0, Standard Error of Mean 1.2 — The adjusted difference from a model may not necessarily match the raw difference between groups

6. Secondary Outcome: AM-PAC-CAT - Daily Activity Domain
Description: as for outcome 4
Time Frame: Baseline to 12-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 6.9 (11.2) | 5.1 (11.3)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.1393, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.7, Standard Error of Mean 1.2; The adjusted difference from a model may not necessarily match the raw difference between groups

7. Secondary Outcome: Accelerometry
Description: Change in lifestyle physical activity will be measured by wrist worn accelerometry to assess change in movement. An index of average total active minutes (≥18mg) per 24 hour period will be prioritized to quantify physical activity volume.
Time Frame: Baseline to 3-month change
Measure: Mean (Standard Deviation); unit: minutes/24 hours
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
minutes/24 hours | 37.3 (95.8) | 13.9 (115.4)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.9257, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.1, Standard Error of Mean 12.3 — The adjusted difference from a model may not necessarily match the raw difference between groups

8. Secondary Outcome: Accelerometry
Description: as for outcome 7
Time Frame: Baseline to 6-month change
Measure: Mean (Standard Deviation); unit: minutes/24 hours
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
minutes/24 hours | 34.0 (100.8) | 18.3 (127.4)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.6588, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.2, Standard Error of Mean 11.8 — The adjusted difference from a model may not necessarily match the raw difference between groups

9. Secondary Outcome: Accelerometry
Description: as for outcome 7
Time Frame: Baseline to 12-month change
Measure: Mean (Standard Deviation); unit: minutes/24 hours
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
minutes/24 hours | 44.8 (121.6) | 12.9 (119.1)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.9920, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 13.0 — The adjusted difference from a model may not necessarily match the raw difference between groups

10. Secondary Outcome: PATIENT HEALTH QUESTIONNAIRE (PHQ-9)
Description: The PHQ-9 is a standardized and validated 9 item depression scale. Scores range from 0-27 points on the scale, with the higher score showing a greater possibility of depression.
Time Frame: Baseline to 3-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | -2.1 (3.1) | -2.2 (2.9)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.9504, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.0, Standard Error of Mean 0.3 — The adjusted difference from a model may not necessarily match the raw difference between groups

11. Secondary Outcome: PATIENT HEALTH QUESTIONNAIRE (PHQ-9)
Description: as for outcome 10
Time Frame: Baseline to 6-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | -1.9 (3.5) | -2.2 (2.8)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.6228, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.2, Standard Error of Mean 0.3 — The adjusted difference from a model may not necessarily match the raw difference between groups

12. Secondary Outcome: PATIENT HEALTH QUESTIONNAIRE (PHQ-9)
Description: as for outcome 10
Time Frame: Baseline to 12-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | -1.7 (3.0) | -2.3 (3.0)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.7966, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.1, Standard Error of Mean 0.3 — The adjusted difference from a model may not necessarily match the raw difference between groups

13. Secondary Outcome: Morley Frail Scale
Description: The Frail Scale is a 5-item assessment of fatigue, resistance, ambulation, illnesses, and loss of weight. Scores range from 0-5 with a higher number indicating greater frailty.
Time Frame: Baseline to 3-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | -0.5 (1.3) | -0.4 (1.3)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.5071, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.1 — The adjusted difference from a model may not necessarily match the raw difference between groups

14. Secondary Outcome: Morley Frail Scale
Description: as for outcome 13
Time Frame: Baseline to 6-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | -0.4 (1.3) | -0.5 (1.4)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.5553, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.1, Standard Error of Mean 0.1 — The adjusted difference from a model may not necessarily match the raw difference between groups

15. Secondary Outcome: Morley Frail Scale
Description: as for outcome 13
Time Frame: Baseline to 12-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | -0.6 (1.3) | -0.4 (1.5)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.1194, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, Standard Error of Mean 0.1 — The adjusted difference from a model may not necessarily match the raw difference between groups

16. Secondary Outcome: Sullivan Cardiac Self-Efficacy
Description: The Sullivan Cardiac Self-Efficacy scale evaluates an individuals confidence to take care of themselves in association to their cardiac disease. It is scored on scale of 0 to 52 points, with a higher score indicating higher confidence.
Time Frame: Baseline to 3-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 3.2 (7.8) | 3.0 (7.9)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.9012, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.8 — The adjusted difference from a model may not necessarily match the raw difference between groups

17. Secondary Outcome: Sullivan Cardiac Self-Efficacy
Description: as for outcome 16
Time Frame: Baseline to 6-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 2.9 (8.9) | 1.8 (8.7)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.4279, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.7, Standard Error of Mean 0.9 — The adjusted difference from a model may not necessarily match the raw difference between groups

18. Secondary Outcome: Sullivan Cardiac Self-Efficacy
Description: as for outcome 16
Time Frame: Baseline to 12-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 2.7 (8.5) | 1.3 (8.7)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.1932, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.1, Standard Error of Mean 0.8 — The adjusted difference from a model may not necessarily match the raw difference between groups

19. Secondary Outcome: THE VETERANS RAND 12-ITEM HEALTH SURVEY (RAND-12) - Physical Component Score
Description: The Veterans RAND-12 is a short standardized and validated questionnaire evaluating quality of life. The 12 items are summarized into two scores, a "Physical Health Summary Measure {PCS-physical component score}" and a "Mental Health Summary Measure {MCS-mental component score}". Both scores range from 0 to 100 with a population mean of 50. These provide an important contrast between physical and psychological health status. A higher score indicates better physical or mental health, respectively.
Time Frame: Baseline to 3-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 7.4 (10.4) | 5.6 (11.8)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.2723, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.4, Standard Error of Mean 1.2 — The adjusted difference from a model may not necessarily match the raw difference between groups

20. Secondary Outcome: THE VETERANS RAND 12-ITEM HEALTH SURVEY (RAND-12) - Physical Component Score
Description: as for outcome 19
Time Frame: Baseline to 6-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 7.1 (10.8) | 7.0 (11.1)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.8951, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.2, Standard Error of Mean 1.2 — The adjusted difference from a model may not necessarily match the raw difference between groups

21. Secondary Outcome: THE VETERANS RAND 12-ITEM HEALTH SURVEY (RAND-12) - Physical Component Score
Description: as for outcome 19
Time Frame: Baseline to 12-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 7.4 (11.6) | 5.1 (13.5)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.2574, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.3, Standard Error of Mean 1.2 — The adjusted difference from a model may not necessarily match the raw difference between groups

22. Secondary Outcome: THE VETERANS RAND 12-ITEM HEALTH SURVEY (RAND-12) - Mental Component Score
Description: RAND-12 is a short questionnaire evaluating quality of life. The 12 items are summarized into two scores, a "Physical Health Summary Measure {PCS-physical component score}" and a "Mental Health Summary Measure {MCS-mental component score}". These provide an important contrast between physical and psychological health status.
Time Frame: Baseline to 3-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 4.6 (9.5) | 5.5 (9.2)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.8307, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, Standard Error of Mean 1.0 — The adjusted difference from a model may not necessarily match the raw difference between groups

23. Secondary Outcome: THE VETERANS RAND 12-ITEM HEALTH SURVEY (RAND-12) - Mental Component Score
Description: as for outcome 22
Time Frame: Baseline to 6-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 4.6 (9.5) | 5.5 (9.2)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.6140, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.5, Standard Error of Mean 1.0 — The adjusted difference from a model may not necessarily match the raw difference between groups

24. Secondary Outcome: THE VETERANS RAND 12-ITEM HEALTH SURVEY (RAND-12) - Mental Component Score
Description: as for outcome 22
Time Frame: Baseline to 12-month change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 4.6 (10.4) | 6.4 (8.2)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.7327, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.3, Standard Error of Mean 1.0 — The adjusted difference from a model may not necessarily match the raw difference between groups

25. Secondary Outcome: Cardiac Rehabilitation Participation
Description: Participants will be asked about participation and adherence in cardiac rehabilitation as well as participants' medical records to evaluate utilization of cardiac rehab. Participation is measured as the number of sessions attended which ranges from 0 to 36. It is assumed that more sessions attended is better.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: number of sessions attended
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
number of sessions attended | 10.1 (12.0) | 10.6 (12.6)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.7651, Wilcoxon rank sum

26. Secondary Outcome: Hospitalizations
Description: Participants will be asked about hospitalizations during blinded monthly calls and follow-up assessments. Participants' medical records may also be reviewed to evaluate readmission to the hospital. Rate of hospitalizations per person year will be reported by group. It is assumed that a lower number of hospitalizations is better.
Time Frame: 12 months
Measure: Number; unit: events per person year
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
events per person year | 0.69 | 0.60
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.3974, Negative binomial regression models; Incident Rate Ratio = 1.15, 95% CI 2-sided [0.83 to 1.59]

27. Secondary Outcome: Duke Activity Status Index (DASI)
Description: The Duke Activity Status Index (DASI) is a self-reported 12-item scale that has been validated in cardiac patients against peak VO2 and has been demonstrated to be a reliable and responsive tool to quantify physical activity in daily living. Scaled scores range from 0 to 58.2 points, with a higher score corresponding to a higher estimated functional capacity.
Time Frame: Baseline to 3-month Change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 10.1 (15.4) | 7.1 (14.2)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.2727, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.7, Standard Error of Mean 1.5 — The adjusted difference from a model may not necessarily match the raw difference between groups

28. Secondary Outcome: Duke Activity Status Index (DASI)
Description: as for outcome 27
Time Frame: Baseline to 6-month Change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 8.5 (15.9) | 7.7 (13.7)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.4269, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.2, Standard Error of Mean 1.5 — The adjusted difference from a model may not necessarily match the raw difference between groups

29. Secondary Outcome: Duke Activity Status Index (DASI)
Description: as for outcome 27
Time Frame: Baseline to 12-month Change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 9.1 (15.6) | 8.0 (15.9)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.4354, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.2, Standard Error of Mean 1.6 — The adjusted difference from a model may not necessarily match the raw difference between groups

30. Secondary Outcome: Rapid Eating Assessment for Participants (Modified REAP-S)
Description: The modified REAP-S is a self-reported 17-item questionnaire used to assess eating habits. The overall summary score ranges from 17 to 53 points, with a higher score representing healthier dietary patterns.
  A modified version of the questionnaire was used for this project after receiving approval by the developers of the instrument.
Time Frame: Baseline to 3-month Change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 2.8 (3.4) | 2.7 (3.9)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.8695, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.4 — The adjusted difference from a model may not necessarily match the raw difference between groups

31. Secondary Outcome: Rapid Eating Assessment for Participants (Modified REAP-S)
Description: as for outcome 30
Time Frame: Baseline to 6-month Change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 3.1 (3.4) | 2.9 (3.8)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.7075, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.4 — The adjusted difference from a model may not necessarily match the raw difference between groups

32. Secondary Outcome: Rapid Eating Assessment for Participants (Modified REAP-S)
Description: as for outcome 30
Time Frame: Baseline to 12-month Change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
score on a scale | 3.1 (3.3) | 3.0 (3.8)
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.8936, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.5 — The adjusted difference from a model may not necessarily match the raw difference between groups

33. Secondary Outcome: Readiness for Change
Description: Interventions like CR that require active engagement by participants are often dependent on the participant's willingness to adopt new activities, habits and routines. The Transtheoretical Model (TTM) is a behavioral framework for understanding readiness for change through 5 change-stages: (1) precontemplation, (2) contemplation, (3) preparation, (4) action, (5) maintenance. Participants in this study are asked at baseline "Are you ready to make some healthy lifestyle changes to help your heart?", and at each follow-up assessment "Since your hospitalization for your heart, have you made or are you making some healthy lifestyle changes to help your heart?" to assess current state of change at each time point. The number of participants in each stage of change will be compared between groups at each timepoint. An increased readiness for change is associated with greater likelihood of goal attainment.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 176 | 174
Participants
  Precontemplation | 4 | 5
  Contemplation | 40 | 43
  Preparation | 60 | 55
  Action | 65 | 70
  Maintenance | 7 | 1
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.2794, Chi-squared

34. Secondary Outcome: Readiness for Change
Description: Interventions like CR that require active engagement by participants are often dependent on the participant's willingness to adopt new activities, habits and routines. The Transtheoretical Model (TTM) is a behavioral framework for understanding readiness for change through 5 change-stages: (1) precontemplation, (2) contemplation, (3) preparation, (4) action, (5) maintenance. Participants in this study are asked at baseline "Are you ready to make some healthy lifestyle changes to help your heart?", and at each follow-up assessment "Since your hospitalization for your heart, have you made or are you making some healthy lifestyle changes to help your heart?" to assess current state of change at each time point. The number of participants in each stage of change will be compared between groups at each timepoint.
Time Frame: 3 Months
Population: 153 participants in the MACRO-I arm and 150 in the Usual Care arm completed the Readiness for Change at the 3 month time point.
Measure: Count of Participants; unit: Participants
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 153 | 150
Participants
  Precontemplation | 2 | 3
  Contemplation | 8 | 8
  Preparation | 9 | 14
  Action | 102 | 88
  Maintenance | 32 | 37
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.6177, Chi-squared

35. Secondary Outcome: Readiness for Change
Description: as for outcome 34
Time Frame: 6 Months
Population: 144 participants in the MACRO-I arm and 137 in the Usual Care arm completed the Readiness for Change at the 6 month assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 144 | 137
Participants
  Precontemplation | 5 | 2
  Contemplation | 5 | 6
  Preparation | 9 | 18
  Action | 51 | 55
  Maintenance | 74 | 56
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.1440, Chi-squared

36. Secondary Outcome: Readiness for Change
Description: as for outcome 34
Time Frame: 12 Months
Population: 137 participants in the MACRO-I arm and 129 in the Usual Care arm completed the Readiness for Change at the 12 month assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 137 | 129
Participants
  Precontemplation | 8 | 2
  Contemplation | 4 | 9
  Preparation | 10 | 12
  Action | 34 | 40
  Maintenance | 81 | 66
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.1122, Chi-squared

37. Secondary Outcome: Fall Assessment
Description: Falls are a common, deleterious, and expensive aspect of aging which may be preventable via the tenets of MACRO such as good transitional care, age-appropriate exercise, and de-prescribing. We will measure falls as follows: at baseline, we will ask, "Have you had any falls in the past 3 months?" In follow-up assessments, we will ask about interim falls, as well as their severity (e.g., if they caused injury).
  For the outcome assessment, the count of participants in each group who reported having at least one fall over the 12 month period following randomization is reported.
Time Frame: 12 months
Population: 158 participants in the MACRO-i arm and 153 in Usual Care completed the fall assessment at follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | MACRO-I | Usual Care
Number analyzed (Participants) | 158 | 153
Participants | 52 | 50
Statistical Analysis 1: Comparison: MACRO-I vs Usual Care; Test type: Superiority; p = 0.9653, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.63 to 1.62]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for all randomized participants over a 1 year follow-up period.
Description: For any fatal SAEs, if a specific cause of death was not available in the medical chart (e.g. due to subject dying outside of the study site hospital system) the CTCAE term was entered as non-specific "death NOS".
Arm/Group | MACRO-I | Usual Care
All-Cause Mortality (participants affected / at risk) | 8/176 | 12/174
Serious Adverse Events (participants affected / at risk) | 74/176 | 70/174
Other Adverse Events (participants affected / at risk) | 103/176 | 93/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MACRO-I (N=176) | Usual Care (N=174)
ANEMIA (Blood and lymphatic system disorders) | 3 | 2
AORTIC VALVE DISEASE (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 4
ATRIAL FLUTTER (Cardiac disorders) | 1 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 4
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 1 | 0
CHEST PAIN - CARDIAC (Cardiac disorders) | 8 | 4
HEART FAILURE (Cardiac disorders) | 10 | 8
MITRAL VALVE DISEASE (Cardiac disorders) | 2 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 5 | 1
RESTRICTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
SINUS BRADYCARDIA (Cardiac disorders) | 2 | 2
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 2
VERTIGO (Ear and labyrinth disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 0
DIARRHEA (Gastrointestinal disorders) | 1 | 0
DUODENAL HEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 | 0
LOWER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1 | 0
UPPER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
DEATH NOS (General disorders) | 1 | 2
EDEMA LIMBS (General disorders) | 1 | 2
FLU LIKE SYMPTOMS (General disorders) | 2 | 1
MULTI-ORGAN FAILURE (General disorders) | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 2
PAIN (General disorders) | 1 | 0
SUDDEN DEATH NOS (General disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 1 | 0
ENDOCARDITIS INFECTIVE (Infections and infestations) | 0 | 1
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 6 | 1
JOINT INFECTION (Infections and infestations) | 1 | 0
LUNG INFECTION (Infections and infestations) | 4 | 0
SEPSIS (Infections and infestations) | 0 | 2
UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1
WOUND INFECTION (Infections and infestations) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 5 | 5
FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPEC (Injury, poisoning and procedural complications) | 1 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 | 0
CARDIAC TROPONIN T INCREASED (Investigations) | 1 | 0
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 | 2
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 0
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
SOFT TISSUE NECROSIS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 0 | 2
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
INTRACRANIAL HEMORRHAGE (Nervous system disorders) | 1 | 0
ISCHEMIA CEREBROVASCULAR (Nervous system disorders) | 1 | 0
PARESTHESIA (Nervous system disorders) | 1 | 0
STROKE (Nervous system disorders) | 3 | 3
SYNCOPE (Nervous system disorders) | 4 | 1
TRANSIENT ISCHEMIC ATTACKS (Nervous system disorders) | 1 | 2
HALLUCINATIONS (Psychiatric disorders) | 1 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 1 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 2
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 | 0
VAGINAL HEMORRHAGE (Reproductive system and breast disorders) | 0 | 1
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 | 5
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 5
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 6 | 10
HEMATOMA (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 2 | 0
LYMPHEDEMA (Vascular disorders) | 1 | 0
PERIPHERAL ISCHEMIA (Vascular disorders) | 1 | 1
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MACRO-I (N=176) | Usual Care (N=174)
ANEMIA (Blood and lymphatic system disorders) | 3 | 2
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 2 | 2
AORTIC VALVE DISEASE (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 4 | 4
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 3 | 1
CHEST PAIN - CARDIAC (Cardiac disorders) | 6 | 7
LEFT VENTRICULAR SYSTOLIC DYSFUNCTION (Cardiac disorders) | 1 | 0
MITRAL VALVE DISEASE (Cardiac disorders) | 0 | 1
SICK SINUS SYNDROME (Cardiac disorders) | 1 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 2 | 1
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
EAR PAIN (Ear and labyrinth disorders) | 1 | 0
MIDDLE EAR INFLAMMATION (Ear and labyrinth disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 2 | 1
HYPERTHYROIDISM (Endocrine disorders) | 0 | 1
BLURRED VISION (Eye disorders) | 0 | 1
CATARACT (Eye disorders) | 5 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 0
COLITIS (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 0
DENTAL CARIES (Gastrointestinal disorders) | 0 | 1
DIARRHEA (Gastrointestinal disorders) | 5 | 2
ESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 0 | 1
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 | 3
HEMORRHOIDS (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 3 | 0
ORAL HEMORRHAGE (Gastrointestinal disorders) | 0 | 1
EDEMA LIMBS (General disorders) | 5 | 7
FATIGUE (General disorders) | 2 | 2
FLU LIKE SYMPTOMS (General disorders) | 8 | 2
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 3
PAIN (General disorders) | 3 | 11
BRONCHIAL INFECTION (Infections and infestations) | 3 | 1
CONJUNCTIVITIS (Infections and infestations) | 1 | 0
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 25 | 28
JOINT INFECTION (Infections and infestations) | 1 | 0
KIDNEY INFECTION (Infections and infestations) | 1 | 1
LUNG INFECTION (Infections and infestations) | 2 | 1
PHARYNGITIS (Infections and infestations) | 0 | 1
RASH PUSTULAR (Infections and infestations) | 1 | 0
RHINITIS INFECTIVE (Infections and infestations) | 1 | 0
SHINGLES (Infections and infestations) | 0 | 2
SINUSITIS (Infections and infestations) | 3 | 1
TOOTH INFECTION (Infections and infestations) | 0 | 1
UPPER RESPIRATORY INFECTION (Infections and infestations) | 5 | 8
URINARY TRACT INFECTION (Infections and infestations) | 6 | 1
BRUISING (Injury, poisoning and procedural complications) | 1 | 1
BURN (Injury, poisoning and procedural complications) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 24 | 20
FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
INJURY TO CAROTID ARTERY (Injury, poisoning and procedural complications) | 1 | 0
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY (Injury, poisoning and procedural complications) | 1 | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
VACCINATION COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 2
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 1 | 0
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 6
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 1 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 2
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 7
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
DIZZINESS (Nervous system disorders) | 3 | 0
HEADACHE (Nervous system disorders) | 0 | 2
MUSCLE WEAKNESS LEFT-SIDED (Nervous system disorders) | 0 | 1
PARESTHESIA (Nervous system disorders) | 0 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 1 | 3
TRANSIENT ISCHEMIC ATTACKS (Nervous system disorders) | 1 | 0
CONFUSION (Psychiatric disorders) | 0 | 1
DEPRESSION (Psychiatric disorders) | 1 | 0
HEMATURIA (Renal and urinary disorders) | 1 | 1
RENAL CALCULI (Renal and urinary disorders) | 1 | 0
URINARY URGENCY (Renal and urinary disorders) | 1 | 0
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 2
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 4 | 8
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 1
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 2
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 1 | 3
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 8 | 8
HEMATOMA (Vascular disorders) | 1 | 2
HYPERTENSION (Vascular disorders) | 2 | 8
HYPOTENSION (Vascular disorders) | 5 | 3
PERIPHERAL ISCHEMIA (Vascular disorders) | 0 | 1
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT03922529/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT03922529/ICF_001.pdf